CLINICAL TRIAL: NCT00570726
Title: Effect of Needle Bleb Revision With Ranibizumab as a Primary Intervention in a Failing Bleb Following Trabeculectomy
Brief Title: Treatment of Failing Blebs With Ranibizumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The New York Eye & Ear Infirmary (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07.10
Record Dates: First submitted 2007-12-09; First posted 2007-12-11 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2007-12

CONDITIONS: Glaucoma, Open-Angle; Failing Bleb Following Trabeculectomy
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ranibizumab (Lucentis)

SUMMARY:
This study was designed to evaluate the efficacy and safety in the use of Ranibizumab, an effective vascular endothelial growth factor (VGEF) inhibitor, in treating patients with a failing bleb, characterized by increased fibrosis and vascularization of the conjuctiva, following trabeculectomy. Six subjects from one site will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 40 years
* Patients with Open-angle Glaucoma who have had trabeculectomy
* Patients determined to have failing bleb with presence of superficial bleb vascularity and IOP increase on 3 successive visits without topical medication
* Patients whose intraocular pressure (IOP) is above goal IOP after suture lysis and digital compression have been attempted

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation.
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Current infection or inflammation in either eye
* Any abnormality preventing reliable applanation tonometry in either eye
* Other non-glaucomatous disease affecting visual field, (pituitary lesions, demyelinating disease, congenital optic nerve anomaly, prior retinal and optic nerve vascular occlusive disease, retinal dystrophy and degeneration, diabetes and HIV and AIDS infection)
* Strabismus, nystagmus, monocular patient
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2000-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Liebmann, MD, Principal Investigator — Robert Ritch, MD, LLC.
Locations (1):
- Glaucoma Associates of New York, New York, New York, United States